CLINICAL TRIAL: NCT03389477
Title: Los Tres Paso Trial: Step One - Neoadjuvant Palbociclib Monotherapy, Step Two - Concurrent Chemoradiation Therapy, and Step Three - Adjuvant Palbociclib Monotherapy in Patients With p16INK4a Negative, HPV-Unrelated Head and Neck Squamous Cell Carcinoma
Brief Title: Los Tres Paso: Neoadjuvant Palbociclib Monotherapy, Concurrent Chemoradiation Therapy, Adjuvant Palbociclib Monotherapy in Patients With p16INK4a Negative, HPV-Unrelated Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201802162
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — palbociclib; Cetuximab; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: 1: palbociclib, 2: Cisplatin & IMRT, 3: palbociclib (Experimental): * Step 1: Neoadjuvant palbociclib monotherapy (125 mg/day, Days 1-21 of a 28-day cycle for two cycles)
  * Step 2: Cisplatin 100 mg/m^2 given on Days 1 and 22 with accelerated IMRT 70 Gy to be administered over 6 weeks
  * Step 3: Adjuvant palbociclib 125 mg/day, days 1-21 of each 28-day cycle for six cycles. Adjuvant palbociclib will begin 16 to 22 weeks following completion of cisplatin & IMRT
  Interventions: Drug: Palbociclib; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Tumor biopsy; Procedure: Peripheral blood draw
- Cohort 2: 1: palbociclib, 2: Cetuximab & IMRT, 3: palbociclib (Experimental): * Step 1: Neoadjuvant palbociclib monotherapy (125 mg/day, Days 1-21 of a 28-day cycle for two cycles)
  * Step 2: Cetuximab given one week before RT and then weekly with accelerated IMRT 70 Gy to be administered over 6 weeks
  * Step 3: Adjuvant palbociclib 125 mg/day, days 1-21 of each 28-day cycle for six cycles. Adjuvant palbociclib will begin 16 to 22 weeks following completion of cetuximab & IMRT
  Interventions: Drug: Palbociclib; Drug: Cetuximab; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Tumor biopsy; Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is an oral drug available as capsules (or as liquid suspension). The capsules should be taken with food
  Other Names: Ibrance; PD 0332991
Drug: Cetuximab — -Cetuximab must not be administered as an IV push or bolus
  Other Names: Erbitux
  Arms: Cohort 2: 1: palbociclib, 2: Cetuximab & IMRT, 3: palbociclib
Drug: Cisplatin — -Patients will receive cisplatin via intravenous (IV) infusion over 60 minutes.
  Other Names: Platinol-AQ; Platinol
  Arms: Cohort 1: 1: palbociclib, 2: Cisplatin & IMRT, 3: palbociclib
Radiation: Intensity-Modulated Radiation Therapy — -Once daily fractions Monday through Friday, with one additional fraction of RT administered on (preferably) Fridays
  Other Names: IMRT
Procedure: Tumor biopsy — * Tumor tissue will be collected at baseline and then after two cycles of neoadjuvant palbociclib monotherapy
  * If the patient has been previously enrolled in Washington University's TAP protocol (head and neck bank, HRPO #201102323), tissue that has been banked may be accessed in lieu of fresh biopsy at baseline.
Procedure: Peripheral blood draw — Baseline and post-treatment

SUMMARY:
The purpose of this study is to evaluate the results of treating patients with HPV-unrelated head and neck squamous cell carcinoma with neoadjuvant single-agent palbociclib, followed by chemoradiation (either cisplatin + IMRT or cetuximab + IMRT depending on patient characteristics), followed by adjuvant single-agent palbociclib.

ELIGIBILITY:
Inclusion Criteria:

* Larynx SCC, hypopharynx SCC, or oral cavity SCC. HPV-unrelated OPSCC [defined as p16INK4a negative by IHC (staining in < 70% of cells) or HPV High Risk (Type 16 or 18) negative by ISH]. P16INK4a positive larynx SCC, hypopharynx SCC, and oral cavity SCC are eligible given the unknown effect of this on the biology of SCC of these subsites.
* Overall Stage III, IVA, or IVB disease per AJCC version 7.0
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* Normal bone marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
* QTc < 500 msec by Fridericia
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 90 days after completion of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Additional Cohort 1 Eligibility Criteria: Patients enrolling to Cohort 1 must meet all of the following criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function defined as:

  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (IULN) and creatinine clearance ≥ 75 mL/min
  * Bilirubin ≤ 1.5 x IULN
  * ALT and AST ≤ 2.5 x IULN

Additional Cohort 2 Eligibility Criteria: Patients enrolling to Cohort 2 must meet at least one of the following criteria:

* ECOG performance status of 2
* Reduced organ function defined as:

  * Creatinine clearance 30-75 mL/min
  * Bilirubin 1.5-2 x IULN
  * ALT and AST 2.5-5 x IULN

Exclusion Criteria:

* Diagnosis of cutaneous, paranasal sinus, salivary, or nasopharynx SCC, or diagnosis of neck nodes with unknown primary.
* Diagnosis of P16/HPV-ISH positive OPSCC.
* Presence of distant metastatic disease.
* Prior systemic therapy for current diagnosis of HNSCC.
* A history of other malignancy ≤ 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or low risk/curatively treated prostate, thyroid, and cervical cancers.
* Currently receiving any other investigational agents.
* Treated within the last 7 days prior to Day 1 of protocol therapy with:

  * Food or drugs that are known to be STRONG CYP3A4 inhibitors (e.g. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, telithromycin, indinavir, ritonavir, nelfinavir, atazanavir, amprenavir, nefazodone, diltiazem, and delavirdine) or inducers (e.g. glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort) [moderate CYP3A4 inhibitors/inducers are okay]
  * Drugs that are known to prolong the QT interval
  * Drugs that are proton pump inhibitors
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib, cisplatin (for Cohort 1), or cetuximab (for Cohort 2).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (e.g. hypocalcemia, hypokalemia, hypomagnesemia).
* History of cirrhosis.
* History of renal or liver transplant.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 28 days of study entry. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment.
* Known HIV-positivity and on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with palbociclib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Rb (retinoblastoma) loss: mutation or homozygous deletion described on genomic sequencing report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2027-04-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Step 1
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Started | 19 | 7
Completed | 18 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Step 2
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Started | 18 | 7
Completed | 16 | 3
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease progression | 1 | 0
Not completed — Death | 0 | 1
Not completed — Poor performance status and nutrition | 0 | 1
Period: Step 3
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Started | 16 | 3
Completed | 11 | 2
Not Completed | 5 | 1
Not completed — Withdrawal after 3 cycles | 0 | 1
Not completed — Still receiving active treatment | 4 | 0
Not completed — Progressive disease after 2 cycles | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib | Total
Number analyzed (Participants) | 19 | 7 | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 72] | 66 [64 to 75] | 63 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 15 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 7 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 16 | 6 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate of Newly Diagnosed p16INK4a Negative, HPV-unrelated HNSCC to Neoadjuvant Palbociclib Monotherapy
Description: * Tumor response rate is defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR) based on RECIST criteria
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 2 cycles (56 days)
Population: The data for Cohort 1 and Cohort 2 were combined as the participants enrolled in both cohorts received the same neoadjuvant palbociclib treatment (125 mg/day Days 1-21 of a 28-day cycle for two cycles) in Step 1.
Measure: Count of Participants; unit: Participants
Groups:
- Step 1 Neoadjuvant Palbociclib for Cohort 1 and Cohort 2: -Step 1: Neoadjuvant palbociclib monotherapy (125 mg/day, Days 1-21 of a 28-day cycle for two cycles)
Arm/Group | Step 1 Neoadjuvant Palbociclib for Cohort 1 and Cohort 2
Number analyzed (Participants) | 26
Participants | 6

2. Secondary Outcome: Combined Local-regional Disease Relapse Risk and Distant Metastases Risk Following Completion of CRT
Description: * Local-regional disease relapse, a binary variable (Yes vs. No). Local-regional disease relapse rate is defined as the proportion of subjects alive who have local-regional progressed disease at 18 months following completion of CRT, stratified by cohorts.
  * Distant metastases, a binary variable (Yes vs. No). Distant metastases rate is defined as the proportion of subjects alive who have distant metastases at 18 months following completion of CRT, stratified by cohorts.
Time Frame: Through 18 months after completion of step 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Number analyzed (Participants) | 18 | 7
Participants
  Local-regional disease relapse | 0 | 2
  Distant metastases | 4 | 1
  Both local-regional disease relapse and distant metastases | 1 | 0

3. Secondary Outcome: Median Progression-free Survival (PFS) (Stratified by Cohort) of Patients Treated With the Three Step Sequence of Palbociclib Monotherapy, CRT, and Adjuvant Palbociclib Monotherapy
Description: -Progression-free survival (PFS), defined as the interval from the start of Step 2 (CRT) to the first documentation of disease progression or death from any cause or the end of follow-up, stratified by cohorts.
Time Frame: Through 5 years after completion of step 2
Reporting Status: Not Posted, anticipated posting 2028-04

4. Secondary Outcome: Progression-free Survival (PFS) of Patients Treated With the Three Step Sequence of Palbociclib Monotherapy, CRT, and Adjuvant Palbociclib Monotherapy
Description: -Progression-free survival (PFS), defined as the days from the start of Step 2 (CRT) to the first documentation of disease progression or death from any cause or the end of follow-up
Time Frame: Through 2 years after completion of step 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Number analyzed (Participants) | 18 | 7
Participants | 13 | 3

5. Secondary Outcome: Median Overall Survival (OS) of Patients Treated With the Three Step Sequence of Palbociclib Monotherapy, CRT, and Adjuvant Palbociclib Monotherapy
Description: -Overall survival (OS), defined as the days from the time of diagnosis to death from any cause or the end of follow-up
Time Frame: Through 5 years after completion of step 2
Reporting Status: Not Posted, anticipated posting 2028-04

6. Secondary Outcome: Overall Survival of Patients Treated With the Three Step Sequence of Palbociclib Monotherapy, CRT, and Adjuvant Palbociclib Monotherapy
Description: -Overall survival (OS), defined as the days from the time of diagnosis to death from any cause or the end of follow-up
Time Frame: Through 2 years after completion of step 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 1: Palbociclib, 2: Cisplatin & IMRT, 3: Palbociclib | Cohort 2: 1: Palbociclib, 2: Cetuximab & IMRT, 3: Palbociclib
Number analyzed (Participants) | 18 | 7
Participants | 16 | 5

7. Secondary Outcome: Change in Genomic Alterations in Tumor Tissue
Description: Tumor genomic alterations at baseline and at relapse will be compared to assess for potential mechanisms of primary or secondary resistance to palbociclib.
Time Frame: At baseline and at time of disease relapse (up to 5 years)
Reporting Status: Not Posted

8. Secondary Outcome: Association Between Baseline Tumor CDKN2A and CCND1 Alterations and Tumor Response to Palbociclib Given Before CRT and Relapse After CRT
Description: Number of participants with altered versus wild-type at baseline will be compared with response.
Time Frame: At baseline and at time of disease relapse (up to 5 years)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) collected for 56 days Step 1. Step 2 Cohort 1 & Cohort 2 collected 6 weeks. Step 3 collected from start of Step 3 through 30 days following the last day of treatment. If a patient went off treatment during Step 1 or Step 2, they were collected for an additional 30 days after treatment. Median AE follow-up 376.5 days (full range 61-486 days). Median all-cause mortality follow-up 596 days (full range 61 days-1573 days).
Description: Serious adverse events and adverse events were not collected during the long term follow-up.
Groups:
- Step 2 Cohort 1 (Cisplatin + IMRT): -Step 2: Cisplatin 100 mg/m^2 given on Days 1 and 22 with accelerated IMRT 70 Gy to be administered over 6 weeks
- Step 2 Cohort 2 (Cetuximab + IMRT): -Step 2: Cetuximab given one week before RT and then weekly with accelerated IMRT 70 Gy to be administered over 6 weeks
- Step 3 Adjuvant Palbociclib for Cohort 1 and Cohort 2: -Step 3: Adjuvant palbociclib 125 mg/day, days 1-21 of each 28-day cycle for six cycles. Adjuvant palbociclib will begin 16 to 22 weeks following completion of cetuximab & IMRT
- Follow-up After Completion of Treatment: -Follow-up after completion of treatment.
Arm/Group | Step 1 Neoadjuvant Palbociclib for Cohort 1 and Cohort 2 | Step 2 Cohort 1 (Cisplatin + IMRT) | Step 2 Cohort 2 (Cetuximab + IMRT) | Step 3 Adjuvant Palbociclib for Cohort 1 and Cohort 2 | Follow-up After Completion of Treatment
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/18 | 1/7 | 0/19 | 8/26
Serious Adverse Events (participants affected / at risk) | 3/26 | 10/18 | 4/7 | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 26/26 | 18/18 | 7/7 | 19/19 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Neoadjuvant Palbociclib for Cohort 1 and Cohort 2 (N=26) | Step 2 Cohort 1 (Cisplatin + IMRT) (N=18) | Step 2 Cohort 2 (Cetuximab + IMRT) (N=7) | Step 3 Adjuvant Palbociclib for Cohort 1 and Cohort 2 (N=19) | Follow-up After Completion of Treatment (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | NA | NA
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA
Fever (General disorders) | 0 | 1 | 1 | NA | NA
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | NA | NA
Tracheitis (Infections and infestations) | 0 | 1 | 0 | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA | NA
Creatinine increased (Investigations) | 1 | 1 | 0 | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | NA | NA
Platelet count decreased (Investigations) | 0 | 1 | 0 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA
Malabsorption (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Delirium (Psychiatric disorders) | 0 | 2 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | NA | NA
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | NA | NA
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Neoadjuvant Palbociclib for Cohort 1 and Cohort 2 (N=26) | Step 2 Cohort 1 (Cisplatin + IMRT) (N=18) | Step 2 Cohort 2 (Cetuximab + IMRT) (N=7) | Step 3 Adjuvant Palbociclib for Cohort 1 and Cohort 2 (N=19) | Follow-up After Completion of Treatment (N=0)
Anemia (Blood and lymphatic system disorders) | 23 | 17 | 6 | 15 | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | NA
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1 | 3 | NA
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 0 | 0 | NA
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | NA
Tinnitus (Ear and labyrinth disorders) | 2 | 2 | 0 | 2 | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | NA
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | NA
Constipation (Gastrointestinal disorders) | 8 | 13 | 3 | 2 | NA
Diarrhea (Gastrointestinal disorders) | 8 | 7 | 1 | 3 | NA
Dry mouth (Gastrointestinal disorders) | 1 | 15 | 5 | 13 | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | NA
Dysphagia (Gastrointestinal disorders) | 19 | 15 | 4 | 10 | NA
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 0 | 0 | 1 | NA
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA
Mucositis oral (Gastrointestinal disorders) | 1 | 11 | 6 | 5 | NA
Nausea (Gastrointestinal disorders) | 9 | 12 | 5 | 4 | NA
Odynophagia (Gastrointestinal disorders) | 4 | 2 | 1 | 2 | NA
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | NA
Vomiting (Gastrointestinal disorders) | 2 | 9 | 3 | 2 | NA
Edema face (General disorders) | 0 | 0 | 0 | 1 | NA
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | NA
Fatigue (General disorders) | 11 | 13 | 6 | 11 | NA
Fever (General disorders) | 0 | 2 | 0 | 2 | NA
Infusion related reaction (General disorders) | 0 | 0 | 1 | 0 | NA
Localized edema (General disorders) | 0 | 0 | 0 | 1 | NA
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | NA
Pain (General disorders) | 1 | 0 | 0 | 0 | NA
Allergic reaction (dressing adhesive) (Immune system disorders) | 0 | 0 | 1 | 0 | NA
Bacteremia (Infections and infestations) | 0 | 1 | 0 | 0 | NA
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | NA
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA
Lip infection (Infections and infestations) | 1 | 0 | 1 | 0 | NA
Skin infection (Infections and infestations) | 0 | 1 | 1 | 2 | NA
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | NA
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | NA
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 15 | 5 | 6 | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0 | 0 | NA
Alanine aminotransferase increased (Investigations) | 2 | 3 | 1 | 1 | NA
Alkaline phosphatase increased (Investigations) | 4 | 4 | 2 | 3 | NA
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 0 | 2 | NA
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | NA
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0 | NA
Creatinine increased (Investigations) | 3 | 9 | 4 | 6 | NA
Hemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | NA
INR increased (Investigations) | 1 | 3 | 0 | 3 | NA
Lymphocyte count decreased (Investigations) | 15 | 17 | 6 | 18 | NA
Neutrophil count decreased (Investigations) | 20 | 12 | 3 | 17 | NA
Platelet count decreased (Investigations) | 12 | 13 | 3 | 10 | NA
Weight loss (Investigations) | 7 | 14 | 4 | 10 | NA
White blood cell decreased (Investigations) | 20 | 17 | 4 | 19 | NA
Anorexia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2 | NA
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 8 | 2 | 3 | NA
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | NA
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 8 | 5 | 1 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 8 | 3 | 0 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 2 | 8 | 3 | 0 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | NA
Hyponatremia (Metabolism and nutrition disorders) | 7 | 10 | 4 | 6 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 5 | 4 | 3 | NA
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 2 | 1 | 0 | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | NA
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | NA
Dysgeusia (Nervous system disorders) | 3 | 11 | 5 | 11 | NA
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | NA
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 2 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 2 | NA
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | NA
Anxiety (Psychiatric disorders) | 5 | 1 | 2 | 2 | NA
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | NA
Depression (Psychiatric disorders) | 0 | 2 | 1 | 1 | NA
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0 | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1 | NA
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | NA
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | NA
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | NA
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | NA
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | NA
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | NA
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 5 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 6 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 17 | 2 | 2 | 5 | NA
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | NA
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 2 | NA
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | NA
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | NA
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 4 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 3 | NA
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 3 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | NA
Pruritus (ocular) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | NA
Rash pustular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | NA
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | NA
Lymphedema (Vascular disorders) | 0 | 2 | 2 | 5 | NA
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03389477/Prot_SAP_000.pdf